CLINICAL TRIAL: NCT04014647
Title: Peri-operative Measurement of NT-proBNP to Predict Outcomes in Patients Undergoing Elective Vascular Surgery
Brief Title: Measurement Of NT-proBNP to Predict Outcomes in Surgery
Acronym: MOBOS
Status: Suspended | Type: Observational
Why Stopped: Study on hold due to COVID-19 research pause
Sponsor: Julie Dawson (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 260029 (34-03-19)
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Vascular Surgical Procedure
Keywords: Vascular Surgical Procedure; Pro-brain natriuretic peptide (1-76); Natriuretic Peptide, Brain; Troponin I; Galectin 3; Biomarkers; Risk

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Event-free: Patients who have had no negative events (as described in group 2)
- Negative event: Group 2 - patients with one or more of the following negative events post-operatively:
  * Whether the patient has been prescribed inotropic support
  * Wound infection by assessing use of antibiotics.
  * Length of stay in hospital >1 week
  * Reduced renal function assessed by having any AKI alert during hospital stay
  * Cardiac event within 31 days following surgery
  * Death within 31 days following surgery

SUMMARY:
The team is investigating whether N-terminal pro B-type natriuretic peptide (NT-proBNP) and other cardiac markers are useful for predicting outcomes for patients undergoing vascular surgery. By measuring NT-proBNP before and after surgery, the investigators may be able to determine which patients are at risk of an adverse outcome, such as a heart attack or death.

DETAILED DESCRIPTION:
Almost 1 in 5 patients who have elective major vascular surgery experience death or a myocardial infarction (MI) at 18 months post-surgery. Research has shown that peri-operative interventions may improve outcomes for high-risk patients. Cardiac bio-markers may be used to identify these high-risk patients, in particular pre- and post-operative NT-proBNP.

Mahla found that by comparing surgery outcomes with NT-proBNP concentrations peri-operatively, high-risk patients could be identified and subsequent therapeutic decisions could be made to minimise adverse outcomes.

Van Kimmenade evaluated patients with acute heart failure and found that galectin-3 (Gal-3) was the best predictor of 60-day mortality compared with NT-proBNP and apelin (another cardiac marker), whereas NT-proBNP was the most useful for diagnosing HF. The authors also found that the combination of both markers (Gal-3 and NT-proBNP) have an even higher predictive value for outcome.

The predictive role of troponin I (cTnI) has been observed in a paper by Bursi et al. (2005) where patients undergoing elective major vascular surgery were stratified using the American College of Cardiology/American Heart Association (ACC/AHA) guidelines and followed up over a period of 24 months. Patients in every group with an elevated post-operative cTnI (≥100ng/L) were at greater risk of either MI or death.

The successful identification of high-risk patients can go on to have interventional risk-reducing pharmacological, therapeutic, diagnostic, or observational measures.

Prevention of cardiovascular events, particular for an aging population, can have positive impact on both the patient and society as a whole as it may result in patients maintaining their independence, avoiding major illness, avoiding nursing home care and living longer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are equal to or over 18 years old
* Patients scheduled to undergo elective surgery for the following procedures:
* Infrainguinal arterial reconstruction
* Aortic aneurysm
* Aorto-bifemoral bypass / or aortic endarterectomy
* Femoro-popliteal bypass
* Femoro-distal bypass
* Femoral endarterectomy
* Femoro-femoral crossover
* Axillo-femoral bypass
* Elective carotid surgery
* Patients having either general or regional anaesthesia for their surgery

Exclusion Criteria:-

* Patients undergoing emergency surgery
* Those who are unable or unwilling to give informed consent
* Patients with unstable coronary syndromes (acute or recent MI with evidence of important ischemic risk by clinical symptoms or stress testing or unstable or severe angina pectoris)
* Patients with decompensated heart failure (new onset shortness of breath and rales together with echocardiographic evidence of cardiac dysfunction or deterioration of chronic heart failure despite heart failure therapy)
* Patients with chronic atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to have vascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP blood test measured on the day of (pre-) vascular surgery | 4 days
  NT-proBNP blood test measured on the day of (pre-) vascular surgery
NT-proBNP blood test measured on the day 4 after (post-) vascular surgery | 4 days
  NT-proBNP blood test measured on the day 4 after (post-) vascular surgery
Change in NT-proBNP peri-operatively | 4 days
  Change in NT-proBNP peri-operatively

SECONDARY OUTCOMES:
Pre-, post-, and peri-operative troponin I | 4 days
  Pre-, post-, and peri-operative troponin I
Pre-, post-, and peri-operative galectin-3 | 4 days
  Pre-, post-, and peri-operative galectin-3
Pre-, post-, and peri-operative CRP | 4 days
  Pre-, post-, and peri-operative CRP
Pre-, post-, and peri-operative creatinine | 4 days
  Pre-, post-, and peri-operative creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Emma Miler, MSc BSc Hons, Principal Investigator — principle investigator
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Augoustides J, Fleisher LA. Advancing perioperative prediction of cardiac risk after vascular surgery: does postoperative N-terminal pro-brain natriuretic peptide do the trick? Anesthesiology. 2007 Jun;106(6):1080-2. doi: 10.1097/01.anes.0000267586.04132.65. No abstract available. PMID 17525578
- [Background] Bursi F, Babuin L, Barbieri A, Politi L, Zennaro M, Grimaldi T, Rumolo A, Gargiulo M, Stella A, Modena MG, Jaffe AS. Vascular surgery patients: perioperative and long-term risk according to the ACC/AHA guidelines, the additive role of post-operative troponin elevation. Eur Heart J. 2005 Nov;26(22):2448-56. doi: 10.1093/eurheartj/ehi430. Epub 2005 Jul 29. PMID 16055493
- [Background] Canavan M, Smyth A, Robinson SM, Gibson I, Costello C, O'Keeffe ST, Walsh T, Mulkerrin EC, O'Donnell MJ. Attitudes to outcomes measured in clinical trials of cardiovascular prevention. QJM. 2016 Jun;109(6):391-7. doi: 10.1093/qjmed/hcv132. Epub 2015 Jul 31. PMID 26231089
- [Background] Feringa HH, Schouten O, Dunkelgrun M, Bax JJ, Boersma E, Elhendy A, de Jonge R, Karagiannis SE, Vidakovic R, Poldermans D. Plasma N-terminal pro-B-type natriuretic peptide as long-term prognostic marker after major vascular surgery. Heart. 2007 Feb;93(2):226-31. doi: 10.1136/hrt.2006.093716. Epub 2006 Aug 16. PMID 16914484
- [Background] Mahla E, Baumann A, Rehak P, Watzinger N, Vicenzi MN, Maier R, Tiesenhausen K, Metzler H, Toller W. N-terminal pro-brain natriuretic peptide identifies patients at high risk for adverse cardiac outcome after vascular surgery. Anesthesiology. 2007 Jun;106(6):1088-95. doi: 10.1097/01.anes.0000267591.34626.b0. PMID 17525582
- [Background] van Kimmenade RR, Januzzi JL Jr, Ellinor PT, Sharma UC, Bakker JA, Low AF, Martinez A, Crijns HJ, MacRae CA, Menheere PP, Pinto YM. Utility of amino-terminal pro-brain natriuretic peptide, galectin-3, and apelin for the evaluation of patients with acute heart failure. J Am Coll Cardiol. 2006 Sep 19;48(6):1217-24. doi: 10.1016/j.jacc.2006.03.061. Epub 2006 Aug 28. PMID 16979009
- [Background] Yeh HM, Lau HP, Lin JM, Sun WZ, Wang MJ, Lai LP. Preoperative plasma N-terminal pro-brain natriuretic peptide as a marker of cardiac risk in patients undergoing elective non-cardiac surgery. Br J Surg. 2005 Aug;92(8):1041-5. doi: 10.1002/bjs.4947. PMID 15997451